CLINICAL TRIAL: NCT02902575
Title: The Safety and Feasibility of Laparoscopic-assisted Gastrectomy for Advanced Gastric Cancer After Neoadjuvant Chemotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fujian Medical University (Other)
Responsible Party: Principal Investigator, Chang-Ming Huang, Prof., Professor, Fujian Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FUGES-05
Record Dates: First submitted 2016-09-11; First posted 2016-09-16 (Estimated); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Stomach Neoplasms
Keywords: Stomach Neoplasms; Laparoscopy; Advanced Gastric Cancer; Neoadjuvant Chemotherapy
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Intervention Model Description: laparoscopic-assisted gastrectomy for advanced Gastric Cancer after neoadjuvant chemotherapy
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Laparoscopic-assisted Gastrectomy (Experimental): Laparoscopic-assisted gastrectomy with D2 lymphadenectomy will be performed for the treatment of patients assigned to this group
  Interventions: Procedure: Laparoscopic-assisted gastrectomy with D2 lymphadenectomy

INTERVENTIONS:
Procedure: Laparoscopic-assisted gastrectomy with D2 lymphadenectomy — After exclusion of T4b, bulky lymph nodes, or distant metastasis case by diagnostic laparoscopy, Laparoscopic-assisted gastrectomy with D2 lymphadenectomy will be performed with curative treated intent.The type of reconstruction will be selected according to the surgeon's experience and anastomotic procedure is performed extracorporeally using a mini-laparotomy

SUMMARY:
The purpose of this study is to explore the safety, feasibility, long-term and oncologicaloutcomes of laparoscopic-assisted gastrectomy for advanced Gastric Cancer after neoadjuvant chemotherapy.

DETAILED DESCRIPTION:
A prospective single-arm study designed to further evaluate laparoscopic-assisted gastrectomy for advanced Gastric Cancer after neoadjuvant chemotherapy will be performed, to evaluate the safety, feasibility, long-term and oncological outcomes. The evaluation parameters are perioperative mobility and mortality, perioperative clinical efficacy, postoperative life quality, immune function and 3-year survival and recurrence rates.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 75 years
* Primary gastric adenocarcinoma (papillary, tubular, mucinous, signet ring cell, or poorly differentiated) confirmed pathologically by endoscopic biopsy
* cT2-4aN+M0 at preoperative evaluation according to the American Joint Committee on Cancer (AJCC) Cancer Staging Manual Seventh Edition
* No distant metastasis is observed. And the spleen, pancreas or other adjacent organs are not involved by the tumor.
* Performance status of 0 or 1 on Eastern Cooperative Oncology Group scale (ECOG)
* American Society of Anesthesiology score (ASA) class I, II, or III
* Written informed consent

Exclusion Criteria:

* Women during pregnancy or breast-feeding
* Severe mental disorder
* History of previous upper abdominal surgery (except laparoscopic cholecystectomy, previous gastrectomy, endoscopic mucosal resection or endoscopic submucosal dissection)
* History of previous gastrectomy, endoscopic mucosal resection or endoscopic submucosal dissection
* History of other malignant disease within past five years
* History of unstable angina or myocardial infarction within past six months
* History of cerebrovascular accident within past six months
* History of continuous systematic administration of corticosteroids within one month
* Requirement of simultaneous surgery for other disease
* Emergency surgery due to complication (bleeding, obstruction or perforation) caused by gastric cancer
* FEV1<50% of predicted values

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
Morbidity | 30 days
  The early postoperative complication are defined as the event observed within 30 days after surgery.Postoperative complications were graded according to the Clavien-Dindo classiﬁcation system

SECONDARY OUTCOMES:
Pathological response | 30 days
  Pathological response grading was performed according to the Becker TRG system
Radiological response | 30 days
  Radiological response and progression were assessed according to RECIST version 1.1
3-year disease free survival rate | 36 months
  3-year disease free survival rate
3-year overall survival rate | 36 months
  3-year overall survival rate
3-year recurrence pattern | 36 months
  Recurrence patterns are classified into five categories at the time of first diagnosis: locoregional, hematogenous, peritoneal, distant lymph node, and mixed type
Mortality | 30 days
  The early mortality are defined as the event observed within 30 days after surgery.
Time to first ambulation | 10 days
  The data of postoperative recovery course
Rates of combined organ resection | 1 day
  Combined organ resection performing by severe injury or abdominal adhesions
The number of lymph node dissection | 1 day
  The number of lymph node dissection
The variation of weight | 12 months
  The variation of weight on postoperative 3, 6, 9 and 12 months
The daily highest body temperature | 7 days
  The daily highest body temperature before discharge
Time to first flatus | 10 days
  Time to first flatus
Time to first liquid diet | 10 days
  Time to first liquid diet
Time to soft diet | 10 days
  Time to soft diet
Scale the amount of abdominal drainage | 10 days
  Scale the amount of abdominal drainage
Blood transfusion | 10 days
  Blood transfusion
The number of positive lymph nodes | 1 days
  The number of positive lymph nodes
Intraoperative lymph node dissection time | 1 days
  intraoperative lymph node dissection time includes infrapyloric area lymph node,suprapancreatic area lymph node,splenic hilar area lymph node, cardial area lymph node and jejunal lymph nodes adjacent to the anastomosis.
Intraoperative blood loss | 1 days
  Intraoperative blood loss
Time of operation | 1 day
  Time of operation
Intraoperative injury | 1 days
  Intraoperative injury
The amount of use of titanium clip | 1 days
  The amount of use of titanium clip
The rate of conversion to laparotomy | 1 days
  The rate of conversion to laparotomy
The variation of albumin | 12 month
  The variation of albumin on postoperative 3, 6, 9 and 12 months
The results of endoscopy | 12 month
  the results of endoscopy on postoperative 3 and 12 months
The values of white blood cell count | 7 days
  the values of white blood cell count from peripheral blood before operation and on postoperative day 1, 3, 5 are recorded
The values of hemoglobin | 7 days
  the values of hemoglobin from peripheral blood before operation and on postoperative day 1, 3, 5 are recorded.
The values of C-reactive protein | 7 days
  the values of C-reactive protein from peripheral blood before operation and on postoperative day 1, 3, 5 are recorded.
The values of prealbumin | 7 days
  the values of prealbumin from peripheral blood before operation and on postoperative day 1, 3, 5 are recorded.
Duration of hospital stay | 10 days
  Duration of hospital stay
Late postoperative complication | 36 months
  The late postoperative complication was defined as the event observed within the period from postoperative day 31th to the end of month 36th.
Adverse events | 30 days
  Adverse events (AEs) of neoadjuvant chemotherapy were assessed at each visit per the National Cancer Institute Common Terminology Criteria for Adverse Events (version 4.0)